CLINICAL TRIAL: NCT01620242
Title: A PHASE II, OPEN-LABEL, MULTICENTER TRIAL OF CABAZITAXEL IN PATIENTS WITH RECURRENT OR METASTATIC HEAD AND NECK CANCER AFTER FAILURE OF CISPLATIN, CETUXIMAB AND TAXANES.
Acronym: ORL03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0130/1106; 2011-004712-32 (EudraCT Number)
Record Dates: First submitted 2012-05-24; First posted 2012-06-15 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Recurrent Head and Neck Cancer; Metastatic Head and Neck Cancer
Keywords: recurrent or metastatic head and neck cancer; cabazitaxel
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): All patients are treated with Cabazitaxel.
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — 25 mg/m2 every 3 weeks by IV administration

SUMMARY:
This is a multi-center phase II study assessing whether cabazitaxel could be efficient for treatment of recurrent or metastatic head and neck cancer after failure of cisplatin, cetuximab and taxanes.

DETAILED DESCRIPTION:
Patients will be treated with intravenous cabazitaxel 25 mg/m2 every 3 weeks (D1=D22) for 6 cycles.

In absence of progression disease or unacceptable toxicity, the treatment could be continued until a maximum of 10 cycles.

Disease response will be assessed every 6 weeks (i.e. every 2 cycles) clinically and by CT-scan.

An interim analysis will be carried out after the inclusion of the first 10 eligible and assessable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or recurrent Head and neck cancer
2. Progression after cisplatin, cetuximab and taxanes (drugs could have been administered alone or in combination) given for recurrent/metastatic disease
3. Age ≥ 18
4. ECOG performance status ≤ 2
5. At least one measurable lesion on CT-scan (as per RECIST criteria V1.1).
6. Life expectancy ≥ 3 months
7. Adequate hematologic function (neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L; Hb ≥ 9.0 g/dL), renal function (clearance creatinine using the CKD-EPI formula (Chronic Kidney Disease Epidemiology group) ≥ 60 mL/min) and hepatic function (serum bilirubin ≤ 1 ULN; AST and ALT ≤ 2.5 x ULN).
8. Potentially reproductive patients must agree to use an effective contraceptive method while on treatment, beginning 2 weeks before the first dose of investigational product and for 6 months after the final dose of investigational product.
9. Women of childbearing potential must have a negative serum beta-HCG pregnancy test within 14 days prior of enrolment and/or urine pregnancy test within 48 hours before the first administration of the study treatment.
10. Patients must be affiliated to a Social Security System.
11. Patient who have received the information sheet and signed the informed consent form.
12. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

1. Active concurrent malignancy
2. Progression in the 3 months after the completion of treatment for localized disease
3. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, such as :

   * infection,
   * cardiac disease such as uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within one year, LVEF > grade 2,
   * current active hepatic or biliary disease (with exception of subjects with Gilbert's syndrome, asymptomatic gallstones, liver metastasis or stable chronic liver disease per investigator assessment),
   * renal disease,
   * active GI tract ulceration, malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Subjects with active, uncontrolled ulcerative colitis are also excluded,
   * severely impaired lung function (spirometry and DLCO 70% or less of normal and O2 saturation of 88% or less at rest on room air).
4. Patients must have recovered of previous toxicity of chemotherapy and must not have toxicity grade > 1 ; grade ≥ 2 for neuropathy and grade ≥ 2 for cutaneous rash after cetuximab (in the CTCAE v4.0)
5. Hypersensitivity to cabazitaxel, to other taxanes, or to any excipients of the formulation including polysorbate 80
6. Pregnant women, women who are likely to become pregnant or are breast-feeding.
7. Patients with significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
8. Patients who received any other investigational drugs within the 14 days prior to the start of cabazitaxel.
9. Patients receiving radiation within 4 weeks prior to the first dose of study drug.
10. Patients already included in another therapeutic trial involving an experimental drug
11. Individual deprived of liberty or placed under the authority of a tutor.
12. Other primary tumors within the previous 3 years
13. Concomitant prohibited treatment. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5. A one week wash-out period is necessary for patients who are already on these treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2014-05-27 (Actual)

PRIMARY OUTCOMES:
non-progression at 6 weeks | 6 weeks
  To assess the efficacy of cabazitaxel in terms of non-progression at 6 weeks for the treatment of recurrent or metastatic head and neck cancer after failure of cisplatin, cetuximab and taxanes.
  Non-progression will be assessed after centralized review of CT-scans.

SECONDARY OUTCOMES:
progression free survival | 1-year
Toxicity according to NCI-CTCAE v4.0 | from the first dose up to 30 days after the last dose
Quality of life evaluated by the QLQ-C30 and H&N35 questionnaire | at the inclusion, at 6 weeks and at the end of treatment

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Oscar Lambret, Lille
  - Centre Léon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared at an individual level, those data will be part of the study database including all enrolled patients.